CLINICAL TRIAL: NCT04343573
Title: A Phase II Randomized Study Assessing the Efficacy of Proton Craniospinal Irradiation (CSI) vs Involved-field Photon Radiation Therapy for Leptomeningeal Metastases From Solid Tumor Malignancies
Brief Title: Proton Craniospinal Radiation Therapy vs. Partial Photon Radiation Therapy for Leptomeningeal Metastasis From Solid Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-117
Record Dates: First submitted 2020-04-10; First posted 2020-04-13 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Leptomeningeal Metastases
Keywords: Proton Craniospinal Irradiation (CSI); Involved-field Photon Radiation Therapy; 20-117
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Intervention Model Description: This is a randomized (2:1) phase II multicenter trial in patients with leptomeningeal metastases from NSCLC and breast cancer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Proton CSI Followed by Standard of Care (NSCLC & Breast) (Experimental): Proton CSI (30Gy [RBE] in 10 fractions) followed by standard of care systemic treatments for leptomeningeal metastases per physician choice.
  Interventions: Radiation: Proton Craniospinal Irradiation (CSI); Other: Neurocognitive Assessment; Other: MDASI-BT and MDASI-SP
- Standard of Care (Experimental): Involved field photon RT including WBRT and/or focal spine RT (30Gy in 10 fractions) followed by standard of care systemic treatments for leptomeningeal metastases per physician choice.
  Interventions: Radiation: Involved-field Photon Radiation Therapy; Other: Neurocognitive Assessment; Other: MDASI-BT and MDASI-SP
- Proton CSI Followed by Standard of Care (Other Solid Tumors) (Other): (Exploratory arm) Patients with solid tumor malignancies other than NSCLC or breast cancer will be enrolled to the exploratory proton CSI arm (Arm C) and will not undergo randomization. Proton CSI (30Gy [RBE] in 10 fractions) followed by standard of care systemic treatments for leptomeningeal metastases per physician choice.
  Interventions: Radiation: Proton Craniospinal Irradiation (CSI); Other: Neurocognitive Assessment; Other: MDASI-BT and MDASI-SP

INTERVENTIONS:
Radiation: Involved-field Photon Radiation Therapy — Involved field photon RT including WBRT and/or focal spine RT (30Gy in 10 fractions)
  Arms: Standard of Care
Radiation: Proton Craniospinal Irradiation (CSI) — Proton CSI (30Gy [RBE] in 10 fractions)
  Arms: Proton CSI Followed by Standard of Care (NSCLC & Breast); Proton CSI Followed by Standard of Care (Other Solid Tumors)
Other: Neurocognitive Assessment — All patients at MSKCC will complete a neurocognitive test battery at study entry (prior to RT), and approximately 3, 6 and 12 months and post -RT. The neurocognitive tests consists of standardized, validated and reliable measures of attention, executive functions, and memory, for which age- and education-matched healthy control published data are available. Patients will also complete self-report mood and fatigue scales at each of the same time points. This testing will only be done at MSKCC. Non-English-speaking patients and pediatric patients are exempt from completing the neurocognitive assessments. Neurocognitive assessments will be performed in person at MSK-Manhattan; an option to perform follow up assessments via telehealth will be available only for patients who are not able to go to Manhattan for these visits.
Other: MDASI-BT and MDASI-SP — Using MDASI-BT and MDASI-SP questionnaires before, weekly during, at 3 months (+/- 4 weeks), 6 months (+/- 4 weeks), 9 months (+/- 4 weeks), and 12 months (+/- 4 weeks) after group assignment, and at CNS disease progression. Only one set needs to be completed. Non-English-speaking patients and pediatric patients are exempt from completing the patient-reported outcomes unless translated PRO assessment forms are available. Questionnaires will be completed via mail, in-person, or online (MSK Engage).
  Other Names: MD Anderson Symptom Inventory for brain tumors; MD Anderson Symptom Inventory for spine tumors

SUMMARY:
The investigators are doing this study to find out whether proton craniospinal radiation therapy (proton CSI) or partial photon radiation therapy is more effective at preventing leptomeningeal metastasis from worsening. The proton CSI targets the entire space containing the CSF, brain, and spinal fluid. The partial photon radiation therapy treats only areas where the patient is having symptoms, such as the entire brain or part of the spine. The investigators also want to find out if proton CSI improves the symptoms patients may be experiencing because of the leptomeningeal metastasis. In addition, the investigators will compare the side effects of proton CSI and partial photon therapy.

Patients undergoing proton beam RT will receive their treatment at the New York Proton Center in New York, NY. As part of the New York Proton Consortium, MSK has contracted for its faculty to treat patients at the New York Proton Center. If it is unfeasible for patients to get treated at NYPC, patients will have the decision to get treated at ProCure in Summerset, NJ.

ELIGIBILITY:
Inclusion Criteria:

* Patient with solid tumor malignancy with leptomeningeal metastases established radiographically and/or through CSF cytology
* Patients who are candidates for radiation therapy for the treatment of leptomeningeal metastases
* Patients of all ages
* KPS ≥ 60 for participants ≥ 16 years old, and Lansky ≥ 60 for participants < 16 years old
* For adult patient, the patient/ legally authorized representative is able to provide informed consent. For pediatric patient, a parent is able to provide informed consent.
* Adequate bone marrow function:

  * Hemoglobin > 8g/dL
  * Absolute neutrophil count >1,000/mm
  * Platelet count > 100,000/mm
* Female subjects must either be of non-reproductive potential (i.e. pediatric patients, OR postmenopausal by history [≥ 60 years old, or with no menses for >1 year without an alternative medical cause], OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test within 2 weeks prior to starting treatment.
* Patient at reproductive potential must agree to practice an effective contraceptive method.

Exclusion Criteria:

* Patient with multiple, serious major neurologic deficits per physician/investigator assessment including encephalopathy
* Patient with extensive systemic disease and without reasonable systemic treatment options
* Patient who is unable to undergo MRI brain and spine with gadolinium contrast
* Previous radiotherapy to the intended treatment site that precludes developing a treatment plan that respects normal tissue tolerances
* Pregnant or lactating women.

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
CNS progression free survival | 2 years
  For Arm A and Arm B, which will be defined as the duration of time from the date of randomization to the time of progression of disease or death, whichever occurs first. The baseline imaging study will be the diagnostic imaging obtained at study entry.

SECONDARY OUTCOMES:
overall survival (OS) (Arm A and Arm B) | 2 years
  will be included in an analysis of overall survival, defined as time from randomization to death.

CONTACTS AND LOCATIONS:
Overall Officials: Divya Yerramilli, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limitedl protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Yang JT, Yerramilli D, Pentsova E, Wolden S, Young RJ, Correa DD, Imber BS, Wijetunga NA, Goglia AG, Zhang Z, Zheng J, Baser R, Bernstein A, Kratochvil L, Xiao J, Hattangadi-Gluth J, Miller AM, Wilcox JA, Betof Warner A, Yu H, Kris MG, Seidman AD, Powell SN, Boire A. Proton Craniospinal Irradiation for Patients With Leptomeningeal Metastasis: A Randomized Clinical Trial. JAMA Oncol. 2025 Nov 1;11(11):1293-1301. doi: 10.1001/jamaoncol.2025.3007. PMID 40906462
- [Derived] Yang JT, Wijetunga NA, Pentsova E, Wolden S, Young RJ, Correa D, Zhang Z, Zheng J, Steckler A, Bucwinska W, Bernstein A, Betof Warner A, Yu H, Kris MG, Seidman AD, Wilcox JA, Malani R, Lin A, DeAngelis LM, Lee NY, Powell SN, Boire A. Randomized Phase II Trial of Proton Craniospinal Irradiation Versus Photon Involved-Field Radiotherapy for Patients With Solid Tumor Leptomeningeal Metastasis. J Clin Oncol. 2022 Nov 20;40(33):3858-3867. doi: 10.1200/JCO.22.01148. Epub 2022 Jul 8. PMID 35802849
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm